CLINICAL TRIAL: NCT01947777
Title: A Phase 1, Open-Label, Single-Sequence, 2-Period Study to Evaluate the Effect of Rifampin (a CYP3A Inducer) on the Pharmacokinetics of IPI-145 in Healthy Subjects
Brief Title: Phase 1 Study in Healthy Subjects to Evaluate the Effect of Rifampin on the Pharmacokinetics of IPI-145
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IPI-145-11
Record Dates: First submitted 2013-09-18; First posted 2013-09-20 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: Phase 1; Healthy subjects; DDI; CYP3A
MeSH Terms: interventions — duvelisib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IPI-145 — 25 mg oral capsule
Drug: Rifampin — 2x 300 mg oral capsule

SUMMARY:
To evaluate the effect of rifampin, a cytochrome P450 3A (CYP3A) inducer, on the pharmacokinetics (PK) of IPI-145; to assess the safety and tolerability of IPI-145 when administered with rifampin in healthy subjects

DETAILED DESCRIPTION:
* In Treatment Period 1, subjects will receive a single 25 mg oral dose of IPI-145
* In Treatment Period 2, on Days 3-9, the same subjects will receive once daily (QD) oral doses of 600 mg rifampin; on Day 9, subjects will receive a single oral dose of 25 mg IPI-145 concomitantly administered with 600 mg of rifampin

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women of non-childbearing potential between 18-50 years of age
* Body Mass Index (BMI): 18.0 - 32.0 kg/m2
* In good health, determined by no clinically significant findings from clinical evaluations
* Provided written informed consent prior to any study specific procedures

Exclusion Criteria:

* Women of childbearing potential
* Evidence of clinically significant medical conditions
* History of gastrointestinal disease or surgery that may affect drug absorption
* Positive or indeterminate Tuberculosis -spot test at screening
* Any active infection at the time of screening or admission
* Consumption of any nutrients known to modulate cytochrome P450 enzyme activity within 14 days prior to administration of study drug, during the study, and until after discharge

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (AUC) of IPI-145 and its metabolite, IPI-656 | Over 48 hours
Pharmacokinetic parameters (Cmax) of IPI-145 and its metabolite, IPI-656 | Over 48 hours
Pharmacokinetic parameters (t1/2) of IPI-145 and its metabolite, IPI-656 | Over 48 hours
Plasma concentrations of IPI-145 and its metabolite, IPI-656 | Over 48 hours

SECONDARY OUTCOMES:
Incidence of adverse events following administration of IPI-145, rifampin, and the combination. | 2 weeks
  Safety Findings

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (1):
- PRA International, Inc, Lenexa, Kansas, United States